CLINICAL TRIAL: NCT00188058
Title: Comparison of Two Strategies for Setting Positive End-Expiratory Pressure in Acute Lung Injury/ Acute Respiratory Distress Syndrome (ExPress Study).
Brief Title: Comparison of 2 Strategies of Adjustment of Mechanical Ventilation in Patients With Acute Respiratory Distress Syndrome
Acronym: ExPress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRC 01 - 02; DGS : 2002 - 0381
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Acute Respiratory Distress Syndrome; Acute Lung Injury
Keywords: Acute respiratory distress syndrome; Positive end-expiratory pressure; Acute lung injury; Mechanical ventilation; Randomized controlled trial
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minimal alveolar distension (Active Comparator): PEEP is set for a total PEEP (PEEP + intrinsic PEEP) between 5 and 9 cm H2O
  Interventions: Device: Setting of positive end-expiratory pressure
- Maximal alveolar distension (Experimental): PEEP is set for a plateau pressure between 28 and 30 cm H20
  Interventions: Device: Setting of positive end-expiratory pressure

INTERVENTIONS:
Device: Setting of positive end-expiratory pressure

SUMMARY:
The aim of this multicenter randomized controlled trial is to compare the impact on mortality of patients mechanically ventilated for acute lung injury or acute respiratory distress syndrome of two strategies for setting end-expiratory pressure.

DETAILED DESCRIPTION:
Most patients suffering from acute lung injury or acute respiratory distress syndrome require mechanical ventilation. In this setting, positive end-expiratory pressure is used to improve arterial oxygenation. While the beneficial effect on clinical outcome of using low tidal volume is clearly proven, the best way to titrate PEEP is not known. Higher PEEP levels may better improve oxygenation and reduce ventilator-induced lung injury by reducing end-expiratory alveolar collapse but may also cause circulatory depression and aggravate lung injury from end-inspiratory overdistension. This trial compares the impact on outcome of two strategies for setting PEEP. In the "minimal alveolar distension" arm, PEEP is set for a total PEEP (PEEP + intrinsic PEEP) between 5 and 9 cm H20). In the "maximal alveolar recruitment" arm, PEEP is set for a plateau pressure between 28 and 30 cm H20. A tidal volume of 6 ml/kg predicted body weight is used in the two arms. The goals for arterial oxygenation and PaCO2 are the same in the two arms.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation through an endotracheal tube
* Bilateral infiltrates consistent with pulmonary edema
* PaO2/FiO2 < 300 mmHg
* No clinical evidence of left atrial hypertension. If measured, pulmonary artery occlusion pressure < 18 mmHg
* Criteria 1, 2 et 3 jointly present for less than 48 hours
* Written informed consent obtained from the patient or surrogate

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Expected duration of mechanical ventilation through an endotracheal tube < 48 hours
* Participation in other trials within the previous 30 days
* Increased intracranial pressure
* Severe chronic respiratory disease
* Morbid obesity (weight > 1kg/cm)
* Sickle cell disease
* Bone marrow transplant or chemotherapy-induced neutropenia
* Extended burns (> 30 % total body surface area)
* Severe chronic liver disease (Child-Pugh score C)
* Pneumothorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 768 (Actual)
Dates: Start 2002-09 (Actual); Primary Completion 2006-01 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Mortality at 28 days | day 28

SECONDARY OUTCOMES:
Mortality at 60 days | day 60
In hospital mortality | day 60
Ventilator free Days through day 28 | day 28
Number of new organ failure before day 28 | day 28
Proportion of patients alive and unassisted breathing at 28 days | day 28
Number of patients with pneumothorax | day 28
Number of days alive between the first positive "potential weanability test" and day 28 | day 28

CONTACTS AND LOCATIONS:
Overall Officials: ALAIN MERCAT, MD, Principal Investigator — University Hospital of Angers
Locations (44):
- France (44):
  - General Hospital of Aix en Provence, Aix-en-Provence
  - South Hospital of Amiens, Amiens
  - University Hospital of Amiens, Amiens
  - University Hospital of Angers, Angers
  - Victor Dupouy Hospital, Argenteuil
  - General Hospital of Arras, Arras
  - Robert Ballanger Hospital, Aulnay-sous-Bois
  - General Hospital of Avignon, Avignon
  - Hospital of Beauvais, Beauvais
  - Saint André Hospital, Bordeaux
  - University Hospital of Bordeaux, Bordeaux
  - Cavale Blanche Hospital, Brest
  - Hospital of Brive, Brivé
  - Henri Mondor Hospital, Créteil
  - Hospital of Dax, Dax
  - Hospital of Dieppe, Dieppe
  - Departemental Hospital, La Roche-sur-Yon
  - Jacques Monod Hospital, Le Havre
  - Le Kremlin Bicetre Hospital, Le Kremlin-Bicêtre
  - Docteur Schaffner Hospital, Lens
  - University Hospital of Claude Huriez, Lille
  - Croix Rousse Hospital, Lyon
  - Bon Secours Hospital, Metz
  - Saint Eloi Hospital, Montpellier
  - Hospital of Nancy, Nancy
  - University Hospital of Hotel Dieu, Nantes
  - University Hospital of Nimes, Nîmes
  - Oloron Sainte Marie Hospital, Oloron-Sainte-Marie
  - Regional Hospital of Orleans, Orléans
  - Bichat Claude Bernard Hospital, Paris
  - University Hospital of Hôtel Dieu, Paris
  - Hospital Group of Pitié - Salpêtrière, Paris
  - Hospital group of Pitié-Salpêtrière, Paris
  - European Hospital of Georges Pompidou, Paris
  - University Hospital of Jean Bernard, Poitiers
  - University Hospital of La Milètrie, Poitiers
  - René Dubos Hospital, Pontoise
  - Charles Nicolle Hospital, Rouen
  - University Hospital of Rouen, Rouen
  - Saint Aubin Les Elbeuf Hospital, Saint-Aubin-lès-Elbeuf
  - University Hospital of Bellevue, Saint-Etienne
  - Hospital of Soissons, Soissons
  - Hautepierre Hospital, Strasbourg
  - Gustave Dron Hospital, Tourcoing

REFERENCES:
- [Result] Mercat A, Richard J, Brochard L. Comparison of two strategies for setting Peep in ALI/ARDS : EsPress Study.Intensive care med, 19th ESICM Annual Congress - Barcelona, Spain, 2006 Sep, Oral presentation 0365
- [Derived] Diehl JL, Coolen N, Faisy C, Osman D, Prat G, Sebbane M, Nieszkowska A, Gervais C, Richard JC, Richecoeur J, Brochard L, Mercat A, Guerot E, Borgel D. Growth-arrest-specific 6 (GAS6) protein in ARDS patients: determination of plasma levels and influence of PEEP setting. Respir Care. 2013 Nov;58(11):1886-91. doi: 10.4187/respcare.02129. Epub 2013 Apr 9. PMID 23571515
- [Derived] Mercat A, Richard JC, Vielle B, Jaber S, Osman D, Diehl JL, Lefrant JY, Prat G, Richecoeur J, Nieszkowska A, Gervais C, Baudot J, Bouadma L, Brochard L; Expiratory Pressure (Express) Study Group. Positive end-expiratory pressure setting in adults with acute lung injury and acute respiratory distress syndrome: a randomized controlled trial. JAMA. 2008 Feb 13;299(6):646-55. doi: 10.1001/jama.299.6.646. PMID 18270353